CLINICAL TRIAL: NCT06585046
Title: The Risk Factors and Prognosis of Hyperglycemia Secondary to Pancreatic Surgery
Brief Title: Pancreatic Surgery and Risk Factors
Status: Completed | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Shanghai Changzheng Hospital, Shanghai Changzheng Hospital
Other Study IDs: NMU-3CDM-2A
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Surgey; Diabetes Mellitus
Keywords: Pancreatic Surgey; Diabetes Mellitus; PCRD; Risk factor
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: pancreatic surgery — patients who did pancreas-related surgery

SUMMARY:
The goal of this observational study is to learn about post-pancreatic surgery diabetes mellitus(PCRD).The main questions it aims to answer are:

1. What are the clinical characteristics of PCRD?
2. What are the related factors for PCRD? All patients with pancreatic surgery have been given standardized treatment fot the condition.

The researchers will summarize the risk factors for PCRD from the PCRD group.

DETAILED DESCRIPTION:
Sponsors retrospectively collected data from patients with pancreatic surgery in Changzheng centers between January 2017 and June 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and <80 years, male or female; 2. Patients who underwent pancreatic resection in pancreaticobiliary surgery since January 2017 3. Those who have previously completed a cohort study in pancreaticobiliary surgery and signed informed consent; 4. Those who have completed and banked serum specimens and pathology specimens in our hospital.

-

Exclusion Criteria:

1. Age <18 years or ≥80 years; 2. Those with preoperative fasting blood glucose ≥5.8 mmol/l or HbA1c ≥6.0% or a history of diabetes; 3. Those with missing relevant data.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with pancreatic surgery in our centre.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of glycaemic disorders（prevalence of diabetes） (postoperative fasting blood glucose/HbA1C) | (within 5 years after surgery)
  The main objective of this study was the incidence of glucose metabolism disorders in patients treated with pancreatic surgery in our centre.

SECONDARY OUTCOMES:
overall survival | within 5 years after surgery
Disease-Free Survival | within 5 years after surgery

IPD SHARING:
Plan to Share IPD: No